CLINICAL TRIAL: NCT01428882
Title: Phase 4, Prospective, Randomized, Double-blinded, Placebo-controlled Study Comparing Propofol vs. Midazolam Plus Propofol for Nonanesthesiologist Targeted Moderate Sedation in Outpatient Colonoscopy
Brief Title: Propofol vs. Midazolam-based Balanced Propofol for Nonanesthesiologist Moderate Sedation in Colonoscopy
Acronym: MIDAPROP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Infante, Javier Molina, M.D. (Individual)
Responsible Party: Principal Investigator, Javier Molina-Infante, MD, Medical Doctor, Infante, Javier Molina, M.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MIDP11
Record Dates: First submitted 2011-09-02; First posted 2011-09-05 (Estimated); Results first posted 2016-05-25 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-04

CONDITIONS: Procedural Sedation
Keywords: Propofol; Midazolam; Moderate sedation; Deep sedation; Colonoscopy
MeSH Terms: interventions — Midazolam; Propofol

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midazolam balanced propofol sedation (Active Comparator): 2 mg midazolam in 2 ml saline midazolam followed by continuous propofol iv infusion
  Interventions: Drug: Midazolam
- Single-agent propofol sedation (Placebo Comparator): 2 ml saline followed by continuous propofol iv infusion
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Midazolam — Midazolam (5 mg/5 mL) 2 mg before standard propofol induction (0.5-1.5 mg/Kg) and boluses-based sedation during colonoscopy, targeted to a moderate sedation level
  Other Names: Not necessary
  Arms: Midazolam balanced propofol sedation
Drug: Propofol — Placebo (normal saline 2 ml) before standard propofol induction (0.5-1.5 mg/Kg) and boluses-based sedation during colonoscopy, targeted to a moderate sedation level
  Other Names: Not necessary
  Arms: Single-agent propofol sedation

SUMMARY:
Nonanesthesiologist administration of propofol for sedation is actually a field of growing interest for endoscopists, as demonstrated by recent American and European guidelines on this issue. Propofol is a hypnotic drug with rapid onset and offset of action. Used as a single agent, it is commonly titrated to deep sedation, whereas balanced propofol sedation (BPS), which combines propofol with small doses of a benzodiazepine and/or an opioid, can be successfully titrated to moderate sedation. However, nonanesthesiologists propofol administration remains controversial on account of the possibility of deep sedation/general anesthesia related adverse events. On the other hand, the use of longer elimination half-life drugs, such as opioids and benzodiazepines, may theoretically prolong sedation and recovery.

Up to date, no study has addressed a head-to-head comparison of both regimens administered by non-anesthesiologists and titrated to moderate sedation.

This study aims to evaluate the impact on propofol sedation of premedication with a fixed dose of midazolam (2 mg)2 minutes before propofol administration targeted to moderate sedation, in terms of depth of sedation, recovery times, safety and satisfaction.

The onset of sedative action of midazolam has been reported to be 1-2.5 minutes and the peak effect of midazolam occurs 8-12 minutes. Taking into account that colonoscopy usually lasts a minimum of 15-20 minutes, our hypothesis is that synergy between propofol and midazolam may increase the depth of sedation through the initial phases of the procedure, diminishing propofol requirements, but not prolonging significantly recovery times.

DETAILED DESCRIPTION:
Justification of the study:

Nonanesthesiologist administration of propofol is controversial owing to deep sedation concerns. One of the latest therapeutic innovations on this issue has been the development of balanced propofol sedation, which consists of adding low doses of opioids or benzodiazepins. Several studies have recently demonstrated that BPS allows successfully moderate sedation, maintains a reversible drug component, reduces the total dose of propofol even by more than 50% without increasing adverse events and maintains high levels of physician and patient satisfaction, even for advanced endoscopic procedure. However, recovery may be prolonged by using midazolam or meperidine as they have a longer elimination half-life than propofol has.

Up to date, nonanesthesiologist administration of propofol and BPS, using either midazolam or fentanyl, for outpatient colonoscopy have been compared in a single non-placebo controlled randomized trial (VanNatta and Rex, 2006). In this study, the authors obtained shorter recovery times with BPS compared to propofol alone, in contrast with the expected on account of pharmacokinetics. These results can be easily understood yet single-agent propofol was titrated to deep sedation, whereas BPS was titrated to moderate sedation.

Therefore, it is necessary to make a randomized, double-blinded, placebo-controlled trial to directly compare both sedation regimens targeted to a similar moderate level of sedation. The results of this study will conclude which should be the first line treatment for moderate sedation in colonoscopy, providing further insight in drug synergy and its impact on the depth of sedation and recovery times

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing elective outpatient colonoscopy

Exclusion Criteria:

* Age less than 18 years
* Allergy to propofol, soybeans, eggs or midazolam
* Chronic intake of benzodiazepines
* History of colorectal surgery
* ASA class IV, short and tick neck, difficult intubation due to inability to open the mouth widely
* Pregnancy
* Refusal, inability or unwillingness to give written consent
* Patients scheduled for advanced therapeutic colonoscopy or for more than one endoscopic procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2011-06; Primary Completion 2011-10 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Javier Molina-Infante, MD, Principal Investigator — Hospital San Pedro de Alcantara, Caceres, Spain
Locations (1):
- Hospital San Pedro de Alcantara, Cáceres, Caceres, Spain

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Cohen LB. Sedation issues in quality colonoscopy. Gastrointest Endosc Clin N Am. 2010 Oct;20(4):615-27. doi: 10.1016/j.giec.2010.07.003. Epub 2010 Aug 21. PMID 20889067
- [Background] Singh H, Poluha W, Cheung M, Choptain N, Baron KI, Taback SP. Propofol for sedation during colonoscopy. Cochrane Database Syst Rev. 2008 Oct 8;2008(4):CD006268. doi: 10.1002/14651858.CD006268.pub2. PMID 18843709
- [Background] Vargo JJ, Cohen LB, Rex DK, Kwo PY. Position statement: nonanesthesiologist administration of propofol for GI endoscopy. Gastrointest Endosc. 2009 Dec;70(6):1053-9. doi: 10.1016/j.gie.2009.07.020. No abstract available. PMID 19962497
- [Background] Dumonceau JM, Riphaus A, Aparicio JR, Beilenhoff U, Knape JT, Ortmann M, Paspatis G, Ponsioen CY, Racz I, Schreiber F, Vilmann P, Wehrmann T, Wientjes C, Walder B; NAAP Task Force Members. European Society of Gastrointestinal Endoscopy, European Society of Gastroenterology and Endoscopy Nurses and Associates, and the European Society of Anaesthesiology Guideline: Non-anesthesiologist administration of propofol for GI endoscopy. Endoscopy. 2010 Nov;42(11):960-74. doi: 10.1055/s-0030-1255728. Epub 2010 Nov 11. PMID 21072716
- [Background] Rex DK, Deenadayalu VP, Eid E, Imperiale TF, Walker JA, Sandhu K, Clarke AC, Hillman LC, Horiuchi A, Cohen LB, Heuss LT, Peter S, Beglinger C, Sinnott JA, Welton T, Rofail M, Subei I, Sleven R, Jordan P, Goff J, Gerstenberger PD, Munnings H, Tagle M, Sipe BW, Wehrmann T, Di Palma JA, Occhipinti KE, Barbi E, Riphaus A, Amann ST, Tohda G, McClellan T, Thueson C, Morse J, Meah N. Endoscopist-directed administration of propofol: a worldwide safety experience. Gastroenterology. 2009 Oct;137(4):1229-37; quiz 1518-9. doi: 10.1053/j.gastro.2009.06.042. Epub 2009 Jun 21. PMID 19549528
- [Background] Cohen LB, Dubovsky AN, Aisenberg J, Miller KM. Propofol for endoscopic sedation: A protocol for safe and effective administration by the gastroenterologist. Gastrointest Endosc. 2003 Nov;58(5):725-32. doi: 10.1016/s0016-5107(03)02010-8. PMID 14595310
- [Background] Cohen LB, Hightower CD, Wood DA, Miller KM, Aisenberg J. Moderate level sedation during endoscopy: a prospective study using low-dose propofol, meperidine/fentanyl, and midazolam. Gastrointest Endosc. 2004 Jun;59(7):795-803. doi: 10.1016/s0016-5107(04)00349-9. PMID 15173791
- [Background] Rex DK, Deenadayalu V, Eid E. Gastroenterologist-directed propofol: an update. Gastrointest Endosc Clin N Am. 2008 Oct;18(4):717-25, ix. doi: 10.1016/j.giec.2008.06.002. PMID 18922410
- [Background] McQuaid KR, Laine L. A systematic review and meta-analysis of randomized, controlled trials of moderate sedation for routine endoscopic procedures. Gastrointest Endosc. 2008 May;67(6):910-23. doi: 10.1016/j.gie.2007.12.046. PMID 18440381
- [Background] Lee CK, Lee SH, Chung IK, Lee TH, Park SH, Kim EO, Lee SH, Kim HS, Kim SJ. Balanced propofol sedation for therapeutic GI endoscopic procedures: a prospective, randomized study. Gastrointest Endosc. 2011 Feb;73(2):206-14. doi: 10.1016/j.gie.2010.09.035. Epub 2010 Dec 18. PMID 21168838
- [Background] Sipe BW, Scheidler M, Baluyut A, Wright B. A prospective safety study of a low-dose propofol sedation protocol for colonoscopy. Clin Gastroenterol Hepatol. 2007 May;5(5):563-6. doi: 10.1016/j.cgh.2007.01.013. PMID 17478345
- [Background] VanNatta ME, Rex DK. Propofol alone titrated to deep sedation versus propofol in combination with opioids and/or benzodiazepines and titrated to moderate sedation for colonoscopy. Am J Gastroenterol. 2006 Oct;101(10):2209-17. doi: 10.1111/j.1572-0241.2006.00760.x. PMID 17032185
- [Background] Rex DK. Review article: moderate sedation for endoscopy: sedation regimens for non-anaesthesiologists. Aliment Pharmacol Ther. 2006 Jul 15;24(2):163-71. doi: 10.1111/j.1365-2036.2006.02986.x. PMID 16842446
- [Background] Paspatis GA, Manolaraki M, Xirouchakis G, Papanikolaou N, Chlouverakis G, Gritzali A. Synergistic sedation with midazolam and propofol versus midazolam and pethidine in colonoscopies: a prospective, randomized study. Am J Gastroenterol. 2002 Aug;97(8):1963-7. doi: 10.1111/j.1572-0241.2002.05908.x. PMID 12190161
- [Background] Cohen LB. Making 1+1=3: improving sedation through drug synergy. Gastrointest Endosc. 2011 Feb;73(2):215-7. doi: 10.1016/j.gie.2010.10.027. No abstract available. PMID 21295634
- [Background] Padmanabhan U, Leslie K, Eer AS, Maruff P, Silbert BS. Early cognitive impairment after sedation for colonoscopy: the effect of adding midazolam and/or fentanyl to propofol. Anesth Analg. 2009 Nov;109(5):1448-55. doi: 10.1213/ane.0b013e3181a6ad31. Epub 2009 Jul 17. PMID 19617584
- [Background] Kerker A, Hardt C, Schlief HE, Dumoulin FL. Combined sedation with midazolam/propofol for gastrointestinal endoscopy in elderly patients. BMC Gastroenterol. 2010 Jan 27;10:11. doi: 10.1186/1471-230X-10-11. PMID 20105314
- [Derived] Molina-Infante J, Duenas-Sadornil C, Mateos-Rodriguez JM, Perez-Gallardo B, Vinagre-Rodriguez G, Hernandez-Alonso M, Fernandez-Bermejo M, Gonzalez-Huix F. Nonanesthesiologist-administered propofol versus midazolam and propofol, titrated to moderate sedation, for colonoscopy: a randomized controlled trial. Dig Dis Sci. 2012 Sep;57(9):2385-93. doi: 10.1007/s10620-012-2222-4. Epub 2012 May 22. PMID 22615015

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Midazolam Balanced Propofol Sedation | Single-agent Propofol Sedation
Started | 67 | 68
Completed | 61 | 58
Not Completed | 6 | 10
Not completed — Lack of Efficacy | 2 | 7
Not completed — Protocol Violation | 4 | 3

BASELINE CHARACTERISTICS:
Population: Patients were similar at baseline without differences regarding age, gender, body mass index, ASA class or indication for colonoscopy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Midazolam Balanced Propofol Sedation | Single-agent Propofol Sedation | Total
Number analyzed (Participants) | 61 | 58 | 119
Age, Continuous [Mean (Full Range); unit: years] | 58 [19 to 80] | 55 [20 to 86] | 56 [19 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 30 | 64
  Male | 27 | 28 | 55
Body Mass Index [Mean (Standard Deviation); unit: Kg/m2] | 25.8 (4.6) | 25.1 (3.5) | 25.4 (4.1)
Educational degree [Number; unit: participants]
  No degree | 14 | 14 | 28
  High school | 5 | 11 | 16
  Technical | 20 | 10 | 30
  College | 11 | 10 | 21
  Graduate degree | 11 | 13 | 24
ASA class [Number; unit: participants] — ASA 1: a normal healthy patient (e.g., Healthy, non-smoking, no or minimal alcohol use) ASA 2: a patient with mild systemic disease (e.g., current smoker, social alcohol drinker, pregnancy, obesity, well-controlled diabetes mellitus or arterial hypertension) ASA 3: Substantive functional limitations in a patient with one or more moderate to severe diseases (e.g., poorly controlled diabetes mellitus or arterial hypertension, chronic obstructive pulmonary disease, morbid obesity, implanted pacemaker, moderate reduction of ejection fraction, patients on scheduled dialysis)
  participants
    ASA 1 | 22 | 31 | 53
    ASA 2 | 32 | 19 | 51
    ASA 3 | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Level of Sedation Throughout the Entire Procedure
Description: Assessment every two minutes of the level of sedation during the endoscopic procedure, rating it as minimal, moderate or deep.
Time Frame: Up to 1 hour after introduction of the colonoscope
Measure: Number; unit: participants
Arm/Group | Midazolam Balanced Propofol Sedation | Single-agent Propofol Sedation
Number analyzed (Participants) | 61 | 58
participants
  Deep sedation at any point | 22 | 9
  Deep sedation at minute 4 | 10 | 1
  Deep sedation at minute 6 | 12 | 2
  Deep sedation at minute 8 | 10 | 3

2. Secondary Outcome: Duration of Recovery After the Endoscopic Procedure
Description: After completion of the procedure, the patient stood in the examination room monitored continuously by a nurse. When patients responded to normal verbal command, they were asked to sit up and were offered a drink. This was considered the early recovery time.
  If they were able to stand unassisted by the bed and had stable hemodynamics parameters (saturation>90 % on room air and blood pressure and heart rate within 20 % of baseline), they were transferred to a locker room accompanied by a relative. The discharge criteria included ability to stand unassisted and tolerate clear liquids once dressed. Once a patient met discharge criteria, they were allowed to leave at their own discretion
Time Frame: Up to 1 hour after colonoscopy
Measure: Mean (Full Range); unit: minutes
Arm/Group | Midazolam Balanced Propofol Sedation | Single-agent Propofol Sedation
Number analyzed (Participants) | 61 | 58
minutes
  Early recovery time | 6.8 [2 to 16] | 5.3 [2 to 13]
  Discharge time | 10.4 [4 to 26] | 9.80 [2 to 30]

3. Secondary Outcome: Rate of Sedation-related Complications During the Procedure and the Recovery Phases
Description: The following events were considered complications of procedural sedation: a decline in oxygen saturation to less than 85 % longer than 30 s after increasing the oxygen flow rate to 5 L/min and transient propofol interruption, a heart rate less than 40 beats per minute and blood pressure less than 80/50 mmHg. Major complications were defined as need for mechanical ventilation or any cardiorespiratory event requiring anaesthesiologist assistance.
Time Frame: Up to two hours, including colonoscopy performance and recovery period
Measure: Number; unit: participants
Arm/Group | Midazolam Balanced Propofol Sedation | Single-agent Propofol Sedation
Number analyzed (Participants) | 61 | 58
participants
  Transient oxygen desaturation | 5 | 5
  Bradycardia | 2 | 1
  Arterial Hypotension | 3 | 2

4. Secondary Outcome: Rate of Patients and Physician Satisfaction With Sedation
Description: Endoscopists and patients rated their satisfaction with sedation in a 10-cm visual analogue scale after discharge.The patients were contacted 24-48 h after the procedure to answer a questionnaire regarding if they remembered scope insertion or scope removal and willingness to repeat it with a similar protocol and rated their satisfaction and pain perception from 0 to 10. This phone survey was done by the nurse specifically making the measurements in the endoscopy room, who was blinded to the sedation regimen.
  For the interpretation of results of the 0-10 point numerical scale, 0 stands for 'extremely dissatisfied with sedation level during the endoscopic procedure', whereas 10 stands for 'extremely satisfied with sedation level during the endoscopic procedure".
Time Frame: Up to 1 hour after colonoscopy for endoscopists and up to 48 hours for patients
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Midazolam Balanced Propofol Sedation | Single-agent Propofol Sedation
Number analyzed (Participants) | 61 | 58
units on a scale
  Endoscopist Satisfaction | 8.9 [1 to 10] | 8.4 [1 to 10]
  Patient Satisfaction | 9.8 [8 to 10] | 9.5 [5 to 10]

ADVERSE EVENTS:
Arm/Group | Midazolam Balanced Propofol Sedation | Single-agent Propofol Sedation
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/58
Other Adverse Events (participants affected / at risk) | 0/61 | 0/58

LIMITATIONS AND CAVEATS:
Single center study. Small sample size. Fixed and relatively high-dose midazolam (2 mg). Lack of distinction between complications related to either pain stimuli or oversedation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No